CLINICAL TRIAL: NCT03449420
Title: Predictability of Thromboelastography Parameters in Severe Post Partum Hemorrhage : a Retrospective Study
Brief Title: Predictability of Thromboelastography Parameters in Severe Post Partum Hemorrhage
Status: Completed | Type: Observational
Sponsor: Hôpital Armand Trousseau (Other)
Responsible Party: Principal Investigator, Pr Isabelle CONSTANT, Head of Anesthesiology Department, Hôpital Armand Trousseau
Other Study IDs: ArmandTrousseau
Record Dates: First submitted 2017-03-30; First posted 2018-02-28 (Actual); Last update posted 2018-02-28 (Actual); Status verified 2018-02

CONDITIONS: Post Partum Hemorrhage
Keywords: thromboelastography
MeSH Terms: conditions — Postpartum Hemorrhage | interventions — Thrombelastography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Post Partum Hemorrhage: Patients presenting with a post partum hemorrhage. A thromboelastography analysis is realized at discretion of the anesthesiologist in charge
  Interventions: Diagnostic Test: thromboelastography

INTERVENTIONS:
Diagnostic Test: thromboelastography — TEG5000® : Kaolin and Functional Fibrinogen tests on native blood sample

SUMMARY:
The aim of the study is to determine if thromboelastography parameters can be predictive of severe post partum hemorrhage.

ELIGIBILITY:
Inclusion Criteria:

* Women presenting with a post partum hemorrhage
* needing sulprostone infusion
* during third trimester of pregnancy

Exclusion Criteria:

* known coagulation disorders

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — pregnant women
Study Population: Women presenting with a post partum hemorrhage
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2012-01 (Actual); Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Calculated blood loss | during the 24 hours after delivery
  Calculated blood loss at 24 hours after delivery (Sum of the volume of blood transfused and the volume of blood loss calculated by the decrease in hematocrit.)

CONTACTS AND LOCATIONS:
Overall Officials: Agnes Rigouzzo, MD, Study Director — Hôpital Armand Trousseau

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rigouzzo A, Louvet N, Favier R, Ore MV, Piana F, Girault L, Farrugia M, Sabourdin N, Constant I. Assessment of Coagulation by Thromboelastography During Ongoing Postpartum Hemorrhage: A Retrospective Cohort Analysis. Anesth Analg. 2020 Feb;130(2):416-425. doi: 10.1213/ANE.0000000000004422. PMID 31567472